CLINICAL TRIAL: NCT01929434
Title: Efficacy of Stem Cell Transplantation Compared to Rehabilitation Treatment of Children With Cerebral Paralysis
Brief Title: Efficacy of Stem Cell Transplantation Compared to Rehabilitation Treatment of Patients With Cerebral Paralysis
Acronym: CP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-05-13 CP III
Record Dates: First submitted 2013-08-20; First posted 2013-08-28 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2015-07

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; cell transplantation; rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rehabilitation (Active Comparator): Patients in the group accept rehabilitation for three weeks in hospital and other eleven months in their home under the guidance of physical therapist.
  Interventions: Other: rehabilitation
- control (No Intervention): Patients receive no professional treatment in hospital or rehabilitation centre.
- stem cell injection (Experimental): Patients in the group accept cell therapy including four times stem cells transplant via intrathecal injection.
  Interventions: Biological: stem cell injection

INTERVENTIONS:
Other: rehabilitation — Patients only receive rehabilitation of physical therapy and occupational therapy.
  Other Names: phsical exercise rehabilitation
  Arms: rehabilitation
Biological: stem cell injection — Mesenchymal stem cells derived from umbilical cord are transplanted directly into subarachnoid by Lumbar puncture.
  Arms: stem cell injection

SUMMARY:
Cerebral palsy (CP) is described as a group of permanent disorders affecting motor development and posture, resulting in activity limitation attributed to nonprogressive disturbances of the fetal or infant brain. The prevalence of cerebral palsy has increased among the children with low birth-weight, jaundice, respiratory distress and intrauterine infection and so on. The incidence of cerebral palsy is increasing gradually with increased neonatal survival rate. Although there are many kinds of functional therapy programs especially the rehabilitation treatment for cerebral palsy, their effects are limited. Increasing cerebral palsy patients become a heavy burden to the family and society. Stem cell based therapy, a new prospective therapy for central nervous system disorders, has the potential to repair the damaged brain tissue in patients with cerebral palsy.

In this study, 300 patients with cerebral palsy will be divided into three groups and the investigators will use mesenchymal stem cells derived from umbilical cord to treat 100 CP patients of them randomly. We will also follow up the other 100 patients who only receive rehabilitation treatment and another 100 patients who accept neither stem cell therapy nor rehabilitation treatment. On this basis, as the investigators we can compare the efficacy of cell therapy and rehabilitation treatments for cerebral palsy patients.

Multiple sources of assessment were used to ascertain and classify all cases of cerebral palsy. Particularly the Gross Motor Function Measure (GMFM) as an important valid and reliable outcome measure, has made it possible to evaluate the severity of movement disability，change over time and the effects of clinical interventions. It also will be the primary outcome measure in follow-up analysis of this study.

DETAILED DESCRIPTION:
Patients enrolled in this study need to finish our whole follow-up survey for 12 months, which is carried out by clinical doctors, rehabilitators and epidemiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of cerebral palsy.
* Patients' curator must be able to give voluntary consent.

Exclusion Criteria:

* Intracranial infection.
* Severe respiratory and circulatory system diseases.
* Hematologic malignancies.
* Positive serological tests such as AIDS, hepatitis B virus, hepatitis C virus and syphilis （antigen or antibody）.
* Tumors.
* Genetic and metabolic diseases.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure Score | Change from baseline at 12 monthes after enrollment or transplantation
  Gross Motor Function Measure-88 and Gross Motor Function Measure-66

SECONDARY OUTCOMES:
Routine Blood Test and Biochemical Test | Change from baseline at 12 monthes after enrollment or transplantation
  1. red blood cell
  2. white blood cell
  3. platelet count
  4. glutamic pyruvic transaminase
  5. glutamic oxaloacetic transaminase

OTHER OUTCOMES:
Magnetic resonance imaging （MRI） | Change from baseline at 12 monthes after enrollment or transplantation
  The MRI repots would describe brain tissue especially white matter and malacia.

CONTACTS AND LOCATIONS:
Overall Officials: Yihua An, Doctor, Study Director — the General Hospital of Chinese People's Armed Police Forces
Locations (1):
- General Hospital of Chinese People's Armed Police Forces, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Pharoah PO, Platt MJ, Cooke T. The changing epidemiology of cerebral palsy. Arch Dis Child Fetal Neonatal Ed. 1996 Nov;75(3):F169-73. doi: 10.1136/fn.75.3.f169. PMID 8976681
- [Background] Richards CL, Malouin F. Cerebral palsy: definition, assessment and rehabilitation. Handb Clin Neurol. 2013;111:183-95. doi: 10.1016/B978-0-444-52891-9.00018-X. PMID 23622163
- [Background] Himmelmann K. Epidemiology of cerebral palsy. Handb Clin Neurol. 2013;111:163-7. doi: 10.1016/B978-0-444-52891-9.00015-4. No abstract available. PMID 23622160
- [Background] Reddihough DS, Collins KJ. The epidemiology and causes of cerebral palsy. Aust J Physiother. 2003;49(1):7-12. doi: 10.1016/s0004-9514(14)60183-5. PMID 12600249
- [Background] Rethlefsen SA, Ryan DD, Kay RM. Classification systems in cerebral palsy. Orthop Clin North Am. 2010 Oct;41(4):457-67. doi: 10.1016/j.ocl.2010.06.005. PMID 20868878
- [Background] Lubis MU, Tjipta GD, Marbun MD, Saing B. Cerebral palsy. Paediatr Indones. 1990 Mar-Apr;30(3-4):65-70. PMID 2075008